CLINICAL TRIAL: NCT05375734
Title: Phase II, Single-arm Exploratory Clinical Study of Tislelizumab Combined With Anlotinib in the Treatment of Advanced Pulmonary Pleomorphic Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, xiaoshucheng, physicians, Second Affiliated Hospital of Nanchang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-PSC
Record Dates: First submitted 2022-04-10; First posted 2022-05-17 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Pleomorphic Carcinoma; Immunotherapy; Tislelizumab
MeSH Terms: interventions — tislelizumab; anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment group (Experimental): Tislelizumab combined with Anlotinib Tislelizumab：200 mg，ivgtt，d1，Q3W Anlotinib： 10mg P.O d1-d14, Q3W
  Interventions: Drug: Tislelizumab in combination with anlotinib

INTERVENTIONS:
Drug: Tislelizumab in combination with anlotinib — Tislelizumab：200 mg，ivgtt，d1，Q3W anlotinib： 10mg P.O d1-d14, Q3W

SUMMARY:
Evaluate the efficacy and safety of tislelizumab in combination with anlotinib in patients with stage III and IV PSC .

DETAILED DESCRIPTION:
This is a single-arm, prospective, open phase II clinical study to evaluate the efficacy and safety of tislelizumab in combination with anlotinib in patients with stage III and Stage IV PSC. The primary endpoint of this study was Objective Response Rate (ORR).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in the study and sign informed consent;
2. Male or female patients aged between 18 and 80 years;
3. Patients with stage III or IV pulmonary sarcomatoid carcinoma that has been histologically or cytologically confirmed as inoperable or intolerant to radiotherapy and has at least one measurable lesion (according to RECIST V1.1 criteria);EGFR and ALK driver genes were negative.
4. Previous systemic antitumor therapy ≤2 times;
5. ECOG score: 0,1;
6. Life expectancy ≥12 weeks;
7. The main organs function normally, that is, they meet the following criteria:

1) Blood examination standards should be met (no blood transfusion or blood products, g-CSF or other hematopoietic stimulating factors were used within the first 14 days) :HB ≥90 g/L；ANC ≥1.5×109/L (1500/m3)；PLT ≥100×109/L; 2) Biochemical tests shall meet the following standards:TBIL ≤1.5ULN；TBIL≤3ULN in subjects with liver metastases or with proven/suspected Gilbert's disease; ALT and AST≤2.5ULN, whereas ALT and AST≤5ULN in liver metastases. serum creatinine (Cr) ≤1.5ULN or endogenous creatinine clearance (CrCl) ≥50 mL/min (Cockcroft-Gault formula: CrCl (mL/min) =[(140- age)* body weight (kg)* F]/(SCr(mg/dL)*72).Male F=1, female F=0.85, SCr= serum creatinine) (8) Doppler ultrasound assessment: Left ventricular ejection fraction (LVEF) ≥ normal lower limit (50%); (9) Women of childbearing age must have used a reliable contraceptive method or have performed a pregnancy test (serum or urine) within 7 days prior to enrollment with a negative result and be willing to use an appropriate method of contraception during the trial period and 8 weeks after the last dose of the trial drug.For men, consent is required to use an appropriate method of contraception or to have been surgically sterilized during the trial period and 8 weeks after the last administration of the trial drug.

Exclusion Criteria:

(1) Previous antibodies or drugs targeting immune checkpoint pathways, including but not limited to anti-PD-1, anti-PD-L1 or anti-CTLA-4 antibodies; (2) Treatment with systemic immunomodulators (including but not limited to interferon, interleukin-2, and tumor necrosis factor) within 4 weeks prior to randomization or within 5 half-lives of the drug, whichever is longer (cancer vaccine is allowed as part of previous treatment); (3) Imaging (CT or MRI) showed obvious pulmonary cavernous tumor; (4) History and complications

1. Patients with symptomatic brain metastasis, cancerous meningitis, spinal cord compression, or diseases of the brain or pia meningeal revealed by imaging CT or MRI examination during screening (patients with brain metastasis who had completed treatment 4 weeks before enrollment and had stable symptoms without progression could be enrolled, but were confirmed to have no symptoms of cerebral hemorrhage by craniocerebral MRI, CT or venography evaluation);
2. The patient is participating in other clinical studies (excluding non-interventional studies) or less than 4 weeks after the completion of treatment in the previous clinical study;
3. has had or is currently co-existing with other malignancies within the past 2 years, except for cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor infiltrating basal membrane)];
4. Have an active, known or suspected autoimmune disease, including a history of allogeneic organ transplantation, allogeneic hematopoietic stem cell transplantation, hiv-positive history, or acquired immune deficiency syndrome (AIDS).
5. Randomize patients with any disease requiring systemic treatment with corticosteroids (prednisone >10 mg/ day or equivalent) or other immunosuppressive agents within the first 14 days of treatment.
6. Patients who did not recover to NCI-CTCAE≤1 for adverse reactions related to previous anti-tumor therapy (except hair loss);
7. Suffering from serious cardiovascular diseases: grade ⅱ or above myocardial ischemia or myocardial infarction, poorly controlled arrhythmia;Patients with grade ⅲ ~ ⅳ cardiac insufficiency according to NYHA standard, or left ventricular ejection fraction (LVEF) < 50% as indicated by color doppler echocardiography;
8. A history of interstitial lung disease, non-infectious pneumonia or uncontrolled systemic disease, including diabetes, hypertension, pulmonary fibrosis, acute lung disease, etc.Uncontrolled medium to large serous effusion (including pleural effusion, ascites, pericardial effusion), aggravated chronic obstructive pulmonary disease, and active lung infections and/or acute bacterial or fungal respiratory diseases requiring intravenous antibiotic treatment;
9. A known history of severe hypersensitivity to other monoclonal antibodies;
10. A known history of psychotropic drug abuse, alcoholism or drug abuse;
11. Active hepatitis that cannot be controlled after treatment (HEPATITIS B: HBsAg positive and HBV DNA≥1 x 103 copies /ml;Hepatitis C: HCV RNA positive and abnormal liver function);Co-infection with hepatitis B and c; (5) In the judgment of the researcher, the patient may have other factors that may lead to the termination of the study, such as other serious diseases or serious abnormal laboratory tests, or other factors that may affect the safety of the subjects, or family or social factors that may affect the collection of test data and samples.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-08-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate, ORR | Until the disease progression, an average of 1 year
  ORR will be defined as the proportion of participants with a documented, confirmed complete response or partial response per RECIST v1.1.

SECONDARY OUTCOMES:
Progression-free survival, PFS | rom date of treat until the date of first disease progression or date of death from any cause, whichever came first, assessed up to 2 years
  PFS will be defined as the time from the date of randomization to the date of the first objectively documented tumor progression per RECIST v1.1, or death, whichever occurs first PFS will be defined as the time from the date of randomization to the date of the first objectively documented tumor progression per RECIST v1.1, or death, whichever occurs first PFS will be defined as the time from the date of treatment to the date of the first objectively documented tumor progression per RECIST v1.1, or death, whichever occurs first
Disease Control Rate, DCR | Until the disease progression, an average of 1 year
  defined as the proportion of participants whose best overall response (BOR) is complete response, partial response or stable disease as determined by the IRC based on RECIST v1.1 defined as the proportion of participants whose best overall response (BOR) is complete response, partial response or stable disease as determined by the IRC based on RECIST v1.1
Proportion of adverse events | Up to approximately 12 months or end of treatment visit, whichever came first
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Afiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No